CLINICAL TRIAL: NCT00555048
Title: A Prospective Trial to Evaluate the Role of In Vivo T Cell Depletion by Campath® (Alemtuzumab) in Reduction of Transplant Related Mortality in Transplantation From HLA-Class I or Class II Mismatched, Unrelated Donors
Brief Title: Alemtuzumab, Busulfan, and Cyclophosphamide Followed By a Donor Stem Cell Transplant in Treating Patients With Hematologic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ann Woolfrey, Principal Investigator, Fred Hutchinson Cancer Center
Purpose: Treatment
Other Study IDs: 1981.00; P30CA015704 (NIH); FHCRC-1981.00; CDR0000574145 (Registry Identifier: PDQ)
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Graft Versus Host Disease; Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: graft versus host disease; adult acute megakaryoblastic leukemia (M7); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myelomonocytic leukemia (M4); adult acute promyelocytic leukemia (M3); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); childhood acute megakaryocytic leukemia (M7); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); childhood acute myeloblastic leukemia with maturation (M2); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myelomonocytic leukemia (M4); childhood acute promyelocytic leukemia (M3); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; childhood myelodysplastic syndromes; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative diseases; secondary myelodysplastic syndromes
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Alemtuzumab; Busulfan; Cyclophosphamide; Methotrexate; Tacrolimus; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alemtuzumab (Experimental): Alemtuzumab given together with busulfan and cyclophosphamide followed by a donor stem cell transplant.
  Interventions: Biological: alemtuzumab; Drug: busulfan; Drug: cyclophosphamide; Drug: methotrexate; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: alemtuzumab
Drug: busulfan
Drug: cyclophosphamide
Drug: methotrexate
Drug: tacrolimus
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Monoclonal antibodies, such as alemtuzumab, can find cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Giving chemotherapy drugs, such as busulfan and cyclophosphamide, before a donor stem cell transplant helps stop the growth of cancer cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving tacrolimus and methotrexate after the transplant may stop this from happening.

PURPOSE: This phase I/II trial is studying the best dose of alemtuzumab when given together with busulfan and cyclophosphamide followed by a donor stem cell transplant and to see how well it works in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify the lowest dose of alemtuzumab that is associated with day 180 transplant-related mortality ≤ 45%.

Secondary

* Determine the incidence of life-threatening infection in patients receiving this treatment.
* Determine the incidence of grades III-IV acute graft-vs-host disease (GVHD) in patients receiving this treatment.
* Determine the survival at 1 year in patients receiving this treatment.
* Determine the incidence of disease relapse at 1 year in patients receiving this treatment.
* Determine the incidence of extensive chronic GVHD at 1 year in patients receiving this treatment.
* Determine the incidence of graft failure at day 100 in patients receiving this treatment.

OUTLINE:

* Chemotherapy: Patients receive alemtuzumab IV over 2 hours on days -10 to -6, busulfan IV over 3 hours on days -7 to -4, and cyclophosphamide IV on days -3 and -2.
* Peripheral blood stem cell (PBSC) transplantation: Patients undergo allogeneic filgrastim (G-CSF)-mobilized PBSC transplantation on day 0.
* Graft-vs-host disease prophylaxis: Patients receive tacrolimus IV continuously or orally twice daily on days -1 to 50 and methotrexate IV on days 1, 3, 6, and 11.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of one of the following:

  * Primary acute myeloid leukemia (AML) meeting any of the following criteria:

    * First complete remission (CR; defined as < 5% blasts in marrow) with high-risk features as defined by failure to achieve remission by day 21 after induction chemotherapy, or the presence of chromosomal abnormalities involving any of the following:

      * -5/del(5q)
      * -7/del(7q)
      * Inversion 3q
      * Abnormalities of 11q23, 20q, 21q, del(9q),
      * Translocation 6;9
      * Translocation 9;22
      * Abnormalities of 17p
      * Complex karyotype with ≥ 3 abnormalities
    * Second CR or subsequent in remission
    * Refractory or relapsed disease
  * Secondary AML in remission or relapse
  * Chronic myelogenous leukemia (CML) in accelerated or blast phase meeting the following criteria:

    * Accelerated phase is defined by any one of the following:

      * Blasts 10% to 19% of peripheral blood white cells or bone marrow cells
      * Peripheral blood basophils ≥ 20%
      * Persistent thrombocytopenia (< 100,000/mm³) unrelated to therapy, or persistent thrombocytosis (> 1,000,000/mm³) unresponsive to therapy
      * Increasing spleen size and increasing WBC count unresponsive to therapy
      * Cytogenetic evidence of clonal evolution (i.e., the appearance of an additional genetic abnormality that was not present in the initial specimen at the time of diagnosis of chronic phase CML)
    * Blast phase is defined by any of the following:

      * Blasts ≥ 20% of peripheral blood white cells or bone marrow cells
      * Extramedullary blast proliferation
      * Large foci or clusters of blasts in bone marrow biopsy
  * Primary myelodysplastic syndromes (MDS) with an IPSS score > 1.5
  * Secondary MDS with any IPSS score
  * Primary acute lymphoblastic leukemia meeting any of the following criteria:

    * First CR (< 5% blasts in marrow) with high-risk features as defined by 1 of the following:

      * Failure to achieve remission after first induction chemotherapy
      * Presence of chromosomal abnormalities including hypodiploidy or abnormalities of 11q23 or translocation 9;22
    * Second CR or subsequent in remission
    * Refractory or relapsed disease
* No patients for whom a suitable HLA genotypically identical sibling or fully matched HLA-A, -B, -C, and -DRB1 unrelated donor is available
* No active CNS involvement with disease
* Donors must meet the following criteria:

  * Unrelated volunteer donors who are mismatched for more than one HLA-class I alleles or antigens or for one HLA-class I antigen, but matched by high-resolution typing at HLA-DRB1 and -DQB1, OR who are mismatched for one or more HLA-class II alleles or antigens, but matched by high-resolution typing at HLA-A, -B, and -C

    * No two-antigen mismatch at a single HLA-A, -B, or -C locus
    * No mismatching of class I and class II HLA
    * Matching must be based on results of high-resolution typing at HLA-A, -B, -C, - DRB1, and -DQB1

PATIENT CHARACTERISTICS:

* Karnofsky performance status 50-100%
* No symptomatic coronary artery disease or symptomatic congestive heart failure
* No hepatic disease with transaminases or bilirubin > 2 times upper limit of normal except for isolated hyperbilirubinemia attributed to Gilbert's syndrome
* No severe hypoxemia with room air P_AO_2 < 70, supplemental oxygen-dependence, or DLCO < 60% predicted
* No impaired renal function with creatinine > 2 times upper limit of normal or creatinine clearance < 50% normal
* Not HIV seropositive
* Not pregnant or breast-feeding
* Fertile patients must use effective contraception
* No active infections that are untreated or failing to respond to appropriate therapy

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics

Exclusion criteria:

* Prior allogeneic or autologous bone marrow, peripheral blood stem cell, or umbilical cord blood transplantation using a high-dose total-body irradiation regimen

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2007-09; Primary Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann E. Woolfrey, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Alemtuzumab: Alemtuzumab given together with busulfan and cyclophosphamide followed by a donor stem cell transplant.
  alemtuzumab
  busulfan
  cyclophosphamide
  methotrexate
  tacrolimus
  allogeneic hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
Period: Overall Study
Arm/Group | Alemtuzumab
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 1
Age, Continuous [Median (Full Range); unit: years] | 47 [47 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Lowest Dose of Alemtuzumab Associated With Transplant-related Mortality
Description: Lowest dose of alemtuzumab associated with transplant-related mortality at day 180
Time Frame: Up to day 180
Measure: Number; unit: mg total dose
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 1
mg total dose | 40

2. Secondary Outcome: Life-threatening Infection
Time Frame: Up to 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Grades III-IV Acute Graft-vs-host Disease (GVHD)
Time Frame: Up to 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 1
Participants | 0

4. Secondary Outcome: Overall Survival
Description: Count of surviving participants at 1 year
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 1
Participants | 1

5. Secondary Outcome: Disease Relapse
Description: Count of participants with disease relapse at 1 year
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 1
Participants | 0

6. Secondary Outcome: Extensive Chronic GVHD
Description: Count of participants with extensive chronic GVHD at 1 year
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 1
Participants | 1

7. Secondary Outcome: Graft Failure
Description: Count of participants with graft failure at day 100
Time Frame: Up to day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Arm/Group | Alemtuzumab
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes